CLINICAL TRIAL: NCT01984125
Title: Adolescent Vaccination in the Medical Home
Brief Title: Testing the Use of Prompts to Increase Adolescent Immunization Rates
Acronym: AIMHi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Chief, Division of General Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IP000312
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Vaccine Preventable Diseases; Meningococcal Disease; Human Papillomavirus; Pertussis; Influenza
Keywords: Adolescent Immunization Rates; Provider prompts
MeSH Terms: conditions — Vaccine-Preventable Diseases; Meningococcal Infections; Whooping Cough; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Point-of-Care Prompt (Experimental): A prompt, either electronically or by a nurse, will notify a provider if an adolescent is due for a vaccination. This prompt will appear at any type of visit where the patient is seen by a health provider.
  Interventions: Other: Point-of-Care Prompt
- Control (No Intervention)

INTERVENTIONS:
Other: Point-of-Care Prompt
  Arms: Point-of-Care Prompt

SUMMARY:
Although most US adolescents visit their primary care doctor, their immunization rates are low. Primary care practices from two networks, one in upstate New York as well as a national network of pediatric clinics were surveyed to ask what they thought was the best strategy to increase immunization rates. Point-of-care prompts (either by an electronic health record message or by a nurse) when an adolescent patient comes in for any type of visit and is due for a vaccine was chosen. This study will determine if these prompts will increase immunization rates after a 12-month intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 11 - 18 who had a visit to their primary care provider during the 12 month intervention period

Exclusion Criteria:

* Adolescent is pregnant during intervention time period

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7040 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Adolescent Immunization Rates | One Year
  Bivariate analysis will measure the overall change between the control and intervention groups. Vaccination rates will be summarized using descriptive statistics. As appropriate, two sample t-test or chi-square tests will be used to summarize patient level data. Odds ratio with associated 95% confidence interval will be reported within each of the 2 networks.

SECONDARY OUTCOMES:
Missed Opportunities | One Year
  A hierarchical logistic regression model will evaluate the intervention effect on rates of missed opportunities.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - University of Arkansas - Arkansas Children's Hospital, Little Rock, Arkansas
  - Wilmington Hospital Health Center, Wilmington, Delaware
  - University of Florida, Gainesville, Florida
  - Children's Memorial Hospital - Northwestern University, Chicago, Illinois
  - University of Iowa Hospital, Iowa City, Iowa
  - Boston Children's, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - St. Louis University - School of Medicine, St Louis, Missouri
  - Oak Orchard Community Health Center, Brockport, New York
  - Honeoye Falls Family Medicine, Honeoye Falls, New York
  - Mendon Pediatrics, Mendon, New York
  - Long Pond Pediatrics, Rochester, New York
  - Goodman Pediatrics, Rochester, New York
  - Parkway Pediatrics, Rochester, New York
  - English Road Pediatrics, Rochester, New York
  - 12 Corner Pediatrics, Rochester, New York
  - Westside Pediatrics, Rochester, New York
  - Ridgewood Med-Peds, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Baylor College of Medicine, Texas Children's Hospital, Houston, Texas
  - University of Texas - Houston, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Result] Szilagyi PG, Serwint JR, Humiston SG, Rand CM, Schaffer S, Vincelli P, Dhepyasuwan N, Blumkin A, Albertin C, Curtis CR. Effect of provider prompts on adolescent immunization rates: a randomized trial. Acad Pediatr. 2015 Mar-Apr;15(2):149-57. doi: 10.1016/j.acap.2014.10.006. PMID 25748976